CLINICAL TRIAL: NCT00322673
Title: A Phase 2 Study of XL999 Administered Intravenously to Subjects With Acute Myeloid Leukemia
Brief Title: Study of XL999 in Patients With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to cardiac toxicities
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-207
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Acute Myeloid Leukemia; AML
Keywords: acute myeloid leukemia; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — XL999 was administered at a dose of 2.4 mg/kg given as a 4-hour IV infusion weekly for 4 weeks. In the absence of progressive disease and unacceptable toxicity, subjects were to receive XL999 treatment weekly for up to 1 year on this study

SUMMARY:
This clinical study is being conducted at multiple sites to determine the activity, safety and tolerability of XL999 when given weekly to patients with relapsed or newly-diagnosed AML. XL999 is a small molecule inhibitor against Flk1/kinase insert domain receptor (KDR), PDGFR, c-Kit, FLT3 and SRC. c-Kit and FLT3 are receptors commonly expressed on AML blasts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (except AML FAB-M3 or acute promyelocytic leukemia [APL]) based on the World Health Organization (WHO) classification of ≥ 20% blasts in the bone marrow or peripheral blood at initial diagnosis (prior to start of standard chemotherapy)
* ECOG performance status of 0 or 1
* Subjects with newly-diagnosed AML or subjects with relapsed AML after at least 2 chemotherapy regimens.
* Adequate liver and renal function
* Signed informed consent

Exclusion Criteria:

* Anticancer therapy including chemotherapeutic, biologic, or investigative agents within 30 days of XL999 treatment
* Hematopoietic stem cell transplantation within the previous 6 weeks
* Immunosuppressive therapy (eg, cyclosporine, steroids, tacrolimus) for graft-versus-host disease (GvHD) within 30 days prior to the start of XL999
* The subject has not recovered to grade ≤ 1 or to within 10% of baseline from adverse events due to investigational or chemotherapeutic drugs or stem cell transplantation which were administered > 4 weeks prior to study enrollment
* Uncontrolled and/or concomitant illness
* Pregnant or breastfeeding females
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Hematologic and cytogenetic response rate | Inclusion until disease progression
Safety and tolerability | Inclusion until 30 dyas post last treatment

SECONDARY OUTCOMES:
Duration of hematologic response and transfusion independence | Inclusion until disease progression
Progression-free survival | Inclusion until disease progression
Overall survival | Inclusion until 180-day Follow-up post last treatment or death

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Bui, MD, Study Director — Exelixis
Locations (7):
- United States (7):
  - Eddie Hu, Alhambra, California
  - Ronald Paquette, Los Angeles, California
  - The Thomas and Dorothy Leavey Cancer Center, Northridge, California
  - David Chan, Redondo Beach, California
  - Northwestern University Feinberg School of Medicine, Division of Hematology/Oncology, Chicago, Illinois
  - American Health Network of Indiana, Indianapolis, Indiana
  - Section of Hematology/Oncology Indiana Cancer Pavilion, Indianapolis, Indiana